CLINICAL TRIAL: NCT01661829
Title: A Randomised Controlled Trial for the Effect of Biofeedback Therapy for the Preveintion of Anterior Resection Syndrome in Rectal Cancer Patients Who Have Undergone Low Anterior Resection With Total Mesorectal Excision Following Neoadjuvant Chemoradiation Therapy
Brief Title: An RCT for the Effect of Biofeedback Therapy the Prevention of AR Syndrome in Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kye Bong-Hyeon, Assistant Clinical Professor, The Catholic University of Korea
Other Study IDs: KSVHCRC trial-01; Colorectal disease (Other: Catholic University)
Record Dates: First submitted 2012-08-05; First posted 2012-08-10 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Biofeedback: Patients will undergo biofeedback therapy between 1st adjuvant chemotherapy and stoma closure(= after 3rd ajduvant chemotherapy)
- Kegel: Patients will be trained to take excersise for their anal sphincter by Kegel.

SUMMARY:
In patients who underwent sphincter preserving surgery with toal mesorectal excision and diverting stoma after neoadjuvant chemoradiation therapy for rectal cancer, the inestigators would evaluate the effect of a biofeedback therpy before stoma closure on their anorectal function after stoma closure.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer patients
* neoadjuvant chemoradiation therapy (+)
* sphincter saving surgery with total mesorectal excision (+)
* temporary loop stoma (+)
* adult who is 17 years or older
* patinet who aggree with our study
* if woman is childbearing age, her pregnancy test shoud be indentified 'negative'

Exclusion Criteria:

* patients who have been enrolled to other clinical studies related to this study
* patients who underwent diverting stoma before neoadjuvant chemoradiation
* temporary end -ostomy (+)
* uncontrolled metabolic or systemic disease
* patients who do not understand the purpose of this study because of dementia or pshycologic problem
* MRSA or Clostridium difficille (+)
* Pregnant or during breast feeding
* serious complication after sphincter saving surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients who underwent sphincter saving surgery with total mesorectal excision and diverting stoma after neoadjuvant chemoradiation therapy.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of anterior resection syndrome after stoma closure | 1 year after stoma closure

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colorectal Disease, Department of Surgery, St. Vincent's Hospital, The Catholic University of Korea, Suwon, South Korea

REFERENCES:
- [Derived] Cho HM, Kim H, Yoo R, Kim G, Kye BH. Effect of Biofeedback Therapy during Temporary Stoma Period in Rectal Cancer Patients: A Prospective Randomized Trial. J Clin Med. 2021 Nov 4;10(21):5172. doi: 10.3390/jcm10215172. PMID 34768692
- [Derived] Kye BH, Kim HJ, Kim G, Yoo RN, Cho HM. The Effect of Biofeedback Therapy on Anorectal Function After the Reversal of Temporary Stoma When Administered During the Temporary Stoma Period in Rectal Cancer Patients With Sphincter-Saving Surgery: The Interim Report of a Prospective Randomized Controlled Trial. Medicine (Baltimore). 2016 May;95(18):e3611. doi: 10.1097/MD.0000000000003611. PMID 27149496